CLINICAL TRIAL: NCT01507753
Title: Omega-3 Fatty Acids & Psychoeducational Psychotherapy for Childhood Bipolar Disorder- Not Otherwise Specified
Brief Title: Omega-3 and Therapy Study for Childhood Bipolar Disorder- Not Otherwise Specified
Acronym: OATS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: L. Eugene Arnold (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, L. Eugene Arnold, Principal Investigator, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011H0104; 1R34MH090148-01A1 (NIH)
Record Dates: First submitted 2011-08-12; First posted 2012-01-11 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Bipolar Disorder
Keywords: childhood bipolar disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Supplement and No PEP (Placebo Comparator): Will receive two capsules by mouth, two times daily matched for odor and appearance with the active intervention.
  Interventions: Other: Placebo
- Omega-3 and PEP (Experimental): Omega-3 Supplementation will receive 1000 mg Ω3 (two 500 mg capsules, each containing 350 mg EPA: 50 mg DHA; 100 other Ω3)by mouth, two times daily.
  Psychoeducational Psychotherapy (PEP)Therapy sessions occur twice a week for up to 24 sessions of manualized treatment.
  Interventions: Drug: Omega-3 Supplementation; Behavioral: Psychoeducational Psychotherapy (PEP)
- Omega-3 and No PEP (Experimental): Omega-3 Supplementation will receive 1000 mg Ω3 (two 500 mg capsules, each containing 350 mg EPA: 50 mg DHA; 100 other Ω3)by mouth, two times daily.
  Interventions: Drug: Omega-3 Supplementation
- Placebo Supplement and PEP (Experimental): Placebo Supplement will receive two capsules by mouth, two times daily matched for odor and appearance with the active intervention.
  Psychoeducational Psychotherapy (PEP)Therapy sessions occur twice a week for up to 24 sessions of manualized treatment.
  Interventions: Behavioral: Psychoeducational Psychotherapy (PEP)

INTERVENTIONS:
Drug: Omega-3 Supplementation — The Ω3 group will receive 1000 mg Ω3 (two 500 mg capsules, each containing 350 mg EPA: 50 mg DHA; 100 other Ω3) two times daily for a total daily dose of 2000 mg Ω3 (1400 mg EPA: 200 mg DHA; 400 other Ω3). The placebo group will receive two capsules two times daily matched for odor and appearance with the active intervention.
  Other Names: Omega Brite
  Arms: Omega-3 and No PEP; Omega-3 and PEP
Behavioral: Psychoeducational Psychotherapy (PEP) — Therapy sessions occur twice a week for up to 24 sessions of manualized treatment. The importance of separating symptoms from the individual is emphasized. The family is offered support, validation, and recognition for their own difficult experiences in living with the child's mood disorder. Family members are taught that patients are particularly vulnerable to stress and tension; thus, therapists work with families to reduce the level of stress and tension in their homes. Improvement of communication, problem solving and coping strategies can lead to restoration of hope for recovery and decrease family dysfunction. Goals include strengthening the parent-child bond and helping children and parents feel competent to manage depression now and in future recurrences.
  Other Names: IF-PEP
  Arms: Omega-3 and PEP; Placebo Supplement and PEP
Other: Placebo — The placebo group will receive active monitoring (no IF-PEP) and two capsules two times daily matched for odor and appearance with the active intervention.
  Other Names: Pbo
  Arms: Placebo Supplement and No PEP

SUMMARY:
Childhood bipolar disorder- not otherwise specified (BP-NOS) was originally considered to be a milder version of bipolar disorder (BD). Research now indicates that BP-NOS is a highly impairing condition. No pharmacologic treatment guidelines exist for BP-NOS. Available evidence-based pharmacotherapy guidelines are for BP1; efficacious medications are, unfortunately, associated with significant risk for adverse events (Kowatch et al, 2005; 2009). Previous research on diet and nutrition suggests that omega-3 (Ω3) fatty acids have a beneficial effect on mood, which might provide either a primary or adjunctive treatment with a more favorable risk:benefit ratio for children suffering from BP-NOS than currently available pharmacologic interventions. Psychoeducational psychotherapy (PEP) also has shown promise in treating bipolar spectrum disorders in children aged 8-12 (Fristad, 2006; Fristad, Verducci, Walters, & Young, 2009); its efficacy in treating BP-NOS specifically has not been determined.

The current study compares Ω3, PEP, and their combination to a placebo supplement and active monitoring (AM) in a 12-week trial of 60 children with BP-NOS (15 each with Ω3, Ω3 plus PEP, PEP, and placebo, all with active monitoring). Primary goals are to determine: 1) feasibility of a) recruiting 60 participants in 2 years; b) participant retention over a 12-week trial; and 2) placebo-controlled effect sizes for Ω3, PEP, and combination treatment on manic and depressive symptoms. Secondary goals are to explore response curves over time, mediators and moderators, treatment response across a broad array of outcome variables, adherence to treatment, impact on physiologic parameters often worsened by mood stabilizing medications, and experience of side-effects in participants receiving Ω3 and/or PEP. Comparisons of results to a parallel study of children with depression with identical design will maximize knowledge gained. This pilot study of Ω3, PEP, and combined treatment will provide evidence about whether a larger trial is feasible and justified.

DETAILED DESCRIPTION:
Research indicates BP-NOS is a highly impairing condition comparable to the other bipolar spectrum disorders. Considerable gains have been made recently in understanding BP-NOS, in large part by research utilizing clear operational definitions for BP-NOS. However, clinical trials have focused on youth with Bipolar Disorder- Type I (BP1). No clinical guidelines exist for the treatment of BP-NOS.

No pharmacologic treatment guidelines exist for BP-NOS. Available evidence-based pharmacotherapy guidelines are for BP1 and are associated with significant risk for adverse events. Additionally, while anti-manic agents have been identified, no study has demonstrated an effective anti-depressant agent for youth with bipolar depression. A review of weight gain and metabolic side effects of mood stabilizers and antipsychotic medications in 19 studies of pediatric bipolar patients found significant and clinically relevant weight increases in 18 trials. Clinical trials of depression and bipolar disorders in children and adolescents show approximately 20%-25% of participants dropped out of short-term psychotropic medication treatment trials. Additionally, a recent study of an anticonvulsant mood stabilizer in children failed to show any superiority to placebo.

Previous research on diet and nutrition suggests that omega-3 (Ω3) fatty acids have a beneficial effect on mood with little evidence of negative side-effects or deleterious drug interactions, suggesting Ω3 might function as either a primary or adjunctive treatment with a more favorable risk-benefit ratio for children suffering from BP than currently available pharmacologic interventions.Psychoeducational psychotherapy (PEP) also has shown promise in treating bipolar spectrum disorders in children aged 8-12 its efficacy in treating BP-NOS specifically has not been determined.

The current study compares Ω3, PEP, and their combination to a placebo supplement, all with active monitoring (AM) in a 12-week trial of 60 children with BP-NOS (15 each with Ω3, Ω3 plus PEP, PEP, and placebo. Primary goals are to determine: 1) feasibility of a) recruiting 60 participants in 2 years; b) participant retention over a 12-week trial; and 2) placebo-controlled effect sizes for Ω3, PEP, and combination treatment on manic and depressive symptoms. Secondary goals are to explore response curves over time, mediators and moderators, treatment response across a broad array of outcome variables, adherence to treatment, impact on physiologic parameters often worsened by mood stabilizing medications, and experience of side-effects in participants receiving Ω3 and/or PEP. Comparisons of results to a parallel study of children with depression with identical design will maximize knowledge gained. This pilot study of Ω3, PEP, and combined treatment will provide evidence about whether a larger trial is feasible and justified.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-14 years (boys and girls)
* Has a diagnosis of BP-NOS according to the LAMS definition. Criteria as follows:
* Clinically significant bipolar symptoms that do not meet DSM IV TR criteria for bipolar disorder I or bipolar disorder II
* Elated mood plus 2 or more associated symptoms from DSM IV TR or irritable mood plus 3 or more symptoms
* A change in functioning, and a minimum duration of 4 hours within a 24-hour period and at least 4 cumulative lifetime days meeting criteria
* Full scale IQ ≥ 70
* Child and one parent or other caregiver must be able to complete all assessment
* Child must be able to swallow capsules (training in swallowing will be offered)
* Parent and child must be willing to have blood drawn from child at two study assessments.

Exclusion Criteria:

* Major medical disorders (eg diabetes, epilepsy, metabolic disorder)
* Inability to communicate in English
* Lack of access via phone
* Autism
* Schizophrenia, or other psychotic states warranting anti-psychotic medication
* Active suicidal concern (e.g., "I want to kill myself", a plan for suicide, or an attempt in the past month; however, passive suicidal ideation, such as "I wish I were dead" would not exclude)
* Three or more symptoms rated as "marked" or "severe" on the KDRS or KMRS
* Concurrent mental health intervention (pharmacotherapy and/or psychotherapy) in the past month.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes to K-SADS Mania Rating Scale (KMRS) | Week prior to randomization and then weeks 2, 4, 6, 9, and 12 post-randomization
  This semi-structured interview contains 21 items that assess the severity of manic symptoms in children and adolescents. The KMRS shows high internal consistency (α = 0.94), sensitivity (0.87), and specificity (0.81) (Axelson et al., 2003). The KMRS will be administered at the assessment visits to determine worst lifetime and current (past two weeks) symptoms of mania.

SECONDARY OUTCOMES:
Changes to K-SADS Depression Rating Scale (KDRS) | Week prior to randomization and then weeks 2, 4, 6, 9, and 12 post randomization
  Depressive symptom severity for worst past episode(s) and current episode (past two weeks) will be assessed using the KDRS at the assessment visits. The KDRS is a 12-item semi-structured interview with depression symptoms rated on a 6-point scale from none to severe. The KDRS has been shown to be a reliable measure of symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: L. Eugene Arnold, MD, MEd, Principal Investigator — Ohio State University; Mary A Fristad, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center- Harding Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Vesco AT, Young AS, Arnold LE, Fristad MA. Omega-3 supplementation associated with improved parent-rated executive function in youth with mood disorders: secondary analyses of the omega 3 and therapy (OATS) trials. J Child Psychol Psychiatry. 2018 Jun;59(6):628-636. doi: 10.1111/jcpp.12830. Epub 2017 Oct 24. PMID 29063592
- [Derived] Christian LM, Young AS, Mitchell AM, Belury MA, Gracious BL, Arnold LE, Fristad MA. Body weight affects omega-3 polyunsaturated fatty acid (PUFA) accumulation in youth following supplementation in post-hoc analyses of a randomized controlled trial. PLoS One. 2017 Apr 5;12(4):e0173087. doi: 10.1371/journal.pone.0173087. eCollection 2017. PMID 28379964
- [Derived] Fristad MA, Young AS, Vesco AT, Nader ES, Healy KZ, Gardner W, Wolfson HL, Arnold LE. A Randomized Controlled Trial of Individual Family Psychoeducational Psychotherapy and Omega-3 Fatty Acids in Youth with Subsyndromal Bipolar Disorder. J Child Adolesc Psychopharmacol. 2015 Dec;25(10):764-74. doi: 10.1089/cap.2015.0132. PMID 26682997